CLINICAL TRIAL: NCT01697163
Title: Pilot Study to Identify the Mechanism of De Novo Resistance to Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitors (EGFR-TKIs) in NSCLC With EGFR Mutation.
Brief Title: De Novo Resistance to Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Severance Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Joo Hang Kim, Severance Hospital, Severance Hospital
Other Study IDs: ISSIRES0067
Record Dates: First submitted 2012-09-12; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: NSCLC
Keywords: De Novo Resistance; Iressa; EGFR mutation; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from FFPE tissue sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iressa: Lung cancer patients with EGFR mutation

SUMMARY:
This study is based on the following hypothesis "De novo resistance to EGFR-TKI in EGFR mutation positive patients is related with mutations in EGFR downstream genes".

Investigators will prospectively collect genomic DNA and clinical data regarding treatment outcomes to EGFR-TKI in NSCLC patients with activating EGFR mutations. Investigators will sequence candidate mutations of EGFR downstream genes and analyze c-met gene amplification and protein expression in PTEN, HGF, and IGFR. To identify genetic mutations, amplification, and protein over expression as predictive markers of treatment outcomes, investigators analyzed the association of treatment outcomes with the presence of genetic alteration or protein over expression. Investigators will attempt to identify biomarkers that are able to predict de novo resistance to EGFR-TKI in EGFR mutated NSCLC.

DETAILED DESCRIPTION:
Investigators will prospectively enroll patients who match the following criteria: pathologically proven unresectable NSCLC, planning to treat with EGFR-TKI, patients with activating EGFR mutations, and available tissue sample for DNA extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven unresectable NSCLC
2. 20 years of age or older
3. Planned treatment with Iressa®
4. Patients with activating EGFR mutation (del 19, L858R)
5. Available detailed smoking history
6. Available tissue samples (archival tissue) for mutational or molecular analysis (representative paraffin block or unstained sections from tumor diagnostic specimen are mandatory)
7. Available blood sample
8. At least one lesion that is measurable according to the RECIST 1.1 criteria by CT or MRI
9. Written informed consent

Exclusion Criteria:

1. More than 3rd line treatment
2. Previously treated with other EGFR-TKI
3. Life expectancy of less than 12 weeks
4. Pregnant or lactating female
5. Any unresolved toxicity greater than CTC grade 2 (version 4.0) from previous anti cancer treatment.
6. Unsuitable patient in this treatment as determined by doctor.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patient with EGFR mutation
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
hazard rates of PFS | 1year
  The primary objective is to compare hazard rates of PFS in patients treated with Iressa between with and without any molecular aberrancy in EGFR-downstream genes/proteins.

OTHER OUTCOMES:
OS | 2years
  Overall survival (OS) of EGFR-TKI according to each biomarker (i.e. PIK3CA, AKT, PTEN, and STK11 mutation and HGF, c-met, and IGFR amplification) Disease control rate (DCR) of EGFR-TKI according to each biomarker (i.e. PIK3CA, AKT, PTEN, and STK11 mutation and HGF, c-met, and IGFR amplification) Progression-free survival (PFS) of EGFR-TKI according to each biomarker (i.e. PIK3CA, AKT, PTEN, and STK11 mutation and HGF, c-met, and IGFR amplification)

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hang Kim, MD, PhD, Principal Investigator — Severance Hospital

REFERENCES:
- [Derived] Lim SM, Kim HR, Cho EK, Min YJ, Ahn JS, Ahn MJ, Park K, Cho BC, Lee JH, Jeong HC, Kim EK, Kim JH. Targeted sequencing identifies genetic alterations that confer primary resistance to EGFR tyrosine kinase inhibitor (Korean Lung Cancer Consortium). Oncotarget. 2016 Jun 14;7(24):36311-36320. doi: 10.18632/oncotarget.8904. PMID 27121209